CLINICAL TRIAL: NCT01689532
Title: A Multicenter, Randomized, Double-blind, Parallel Group Study of CNTO 136 (Sirukumab), a Human Anti-IL-6 Monoclonal Antibody, Administered Subcutaneously as Monotherapy, in Japanese Subjects With Active Rheumatoid Arthritis Unresponsive to Methotrexate or Sulfasalazine
Brief Title: A Study of CNTO 136 (Sirukumab) Administered Subcutaneously in Japanese Patients With Active Rheumatoid Arthritis Unresponsive to Methotrexate or Sulfasalazine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR100876; CNTO136ARA3001 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2012-09-18; First posted 2012-09-21 (Estimated); Results first posted 2016-10-27 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-09

CONDITIONS: Arthritis, Rheumatoid
Keywords: Active Rheumatoid Arthritis Unresponsive to Methotrexate or Sulfasalazine; Sirukumab; Human Anti-IL-6 Monoclonal Antibody
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — sirukumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sirukumab 100 mg (Experimental)
  Interventions: Drug: Sirukumab 100 mg
- Sirukumab 50 mg and Placebo (Experimental)
  Interventions: Drug: Sirukumab 50 mg; Drug: Placebo

INTERVENTIONS:
Drug: Sirukumab 100 mg — Sirukumab 100 mg subcutaneous (SC) injection, at Weeks 0, 2, and every 2 weeks through Week 52.
  Arms: Sirukumab 100 mg
Drug: Sirukumab 50 mg — Sirukumab 50 mg SC at Weeks 0, 4, and every 4 weeks through Week 52.
  Arms: Sirukumab 50 mg and Placebo
Drug: Placebo — Between sirukumab injections, placebo SC at Weeks 2, 6, and every 4 weeks through Week 52.
  Arms: Sirukumab 50 mg and Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of sirukumab as a single therapy in Japanese patients with moderately to severely active rheumatoid arthritis (RA) who have not responded to treatment with methotrexate (MTX) or sulfasalazine (SSZ).

DETAILED DESCRIPTION:
This is a randomized (patients will be assigned to treatment by chance), double-blind (study personnel and patients will not know what treatments are being given), multicenter study. The expected duration of the study is 68 weeks. This will include 52 weeks of treatment with study agent with dosing every 2 weeks and 16 weeks of safety follow-up after the last dose. Disease-modifying antirheumatic drugs (DMARDs), including MTX and SSZ, are not permitted from 4 weeks before the first dosing with study agent until Week 24. The use of DMARDs is discouraged at or any time after Week 24; however, patients who have less than 20% improvement from baseline in both swollen and tender joint counts at Week 24 will be allowed to take DMARDs. At or any time after Week 16, the initiation and/or adjustment of oral corticosteroids will be allowed for patients who have less than 20% improvement from baseline in both swollen and tender joint counts at Week 16.

ELIGIBILITY:
Inclusion Criteria:

* Be a Japanese man or woman with a diagnosis of rheumatoid arthritis (RA), according to the revised 1987 criteria of the American Rheumatism Association, for at least 3 months before screening
* Has moderately to severely active RA with at least 6 of 68 tender joints and 6 of 66 swollen joints, at screening and at baseline
* Has been unresponsive to adequate treatment with methotrexate (MTX), sulfasalazine (SSZ), or combination of MTX or SSZ with other disease-modifying antirheumatic drugs (DMARDs) at screening due to lack of benefit after at least 12 weeks of marketed dose of MTX or SSZ, as assessed by the treating physician. Documented lack of benefit may include inadequate improvement in joint counts, physical function, or overall disease activity
* If using oral corticosteroids, must be on a stable dose equivalent to <=10 mg/day of prednisolone for at least 2 weeks prior to first dosing with study agent. If currently not using corticosteroids, the patient must not have received oral corticosteroids (by mouth) for at least 2 weeks prior to first dosing with study agent
* If using nonsteroidal anti-inflammatory drugs (NSAIDs) or other analgesics (pain relievers) for RA, must be on a stable dose for at least 2 weeks prior to first dosing with study agent

Exclusion Criteria:

* Has a history of intolerance to at least 2 or inadequate response to at least one anti-tumor necrosis factor-alpha (anti-TNF-alpha) agent after 3 months of therapy; has received anti-TNF-alpha (eg, infliximab, golimumab, adalimumab, or etanercept) within 3 months of first study agent dosing
* Has a history of intolerance to tocilizumab that precluded further treatment with it, or inadequate response to 3 months of tocilizumab (anti-IL-6 receptor) therapy; has used B-cell-depleting therapy (eg, rituximab) within 7 months of first study agent dosing or has evidence during screening of abnormally low B-cell level caused by previous B-cell depletion therapy; has used any other biologic therapy for the treatment of RA within 3 months of first study agent dosing; has a history of sirukumab use
* Has received intra-articular (IA), intramuscular (IM), or intravenous (IV) corticosteroids for RA, including adrenocorticotrophic hormone during the 4 weeks prior to first study agent dosing
* Has received leflunomide within 24 months before first study agent dosing and has not undergone a drug elimination procedure, unless the M1 metabolite is measured and is undetectable. Drug elimination procedure must be completed prior to obtaining informed consent
* Has a history of cyclophosphamide or cytotoxic agent use; has received cyclosporine A, azathioprine, tacrolimus, mycophenolate mofetil, oral or parenteral gold, or D-penicillamine within 4 weeks of first study agent dosing; has received an investigational drug (including investigational vaccines) or used an investigational medical device within 3 months or 5 half-lives, whichever is longer, before first study agent dosing

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2012-11; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (17):
- Japan (17):
  - Asahikawa
  - Fukuoka
  - Hiroshima
  - Hitachi-Naka
  - Kagoshima
  - Kirishima
  - Kitakyushu
  - Kobe
  - Kumamoto
  - Matsumoto
  - Miyagi
  - Ōita
  - Sapporo
  - Sendai
  - Shizuoka
  - Tokyo
  - Yokohama

REFERENCES:
- [Derived] Takeuchi T, Yamanaka H, Harigai M, Tamamura R, Kato Y, Ukyo Y, Nakano T, Hsu B, Tanaka Y. Sirukumab in rheumatoid arthritis refractory to sulfasalazine or methotrexate: a randomized phase 3 safety and efficacy study in Japanese patients. Arthritis Res Ther. 2018 Mar 7;20(1):42. doi: 10.1186/s13075-018-1536-9. PMID 29514712

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 180 participants who signed informed consent of this study, 122 participants (61 participants in each treatment group) were randomized and treated during the study.
Groups:
- Sirukumab 50 Milligram (mg): Participants received sirukumab 50 milligram (mg) subcutaneous (SC) at Weeks 0, 4, and every 4 weeks (q4w) through Week 52. Between sirukumab injections, participants received placebo SC at Weeks 2, 6, and q4w through Week 52.
- Sirukumab 100 mg: Participants received Sirukumab 100 mg SC at Weeks 0, 2, and every 2 weeks (q2w) through Week 52.
Period: Overall Study
Arm/Group | Sirukumab 50 Milligram (mg) | Sirukumab 100 mg
Started | 61 | 61
Completed | 47 | 52
Not Completed | 14 | 9
Not completed — Adverse Event | 9 | 5
Not completed — Lack of Efficacy | 2 | 2
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Physician Decision | 2 | 0

BASELINE CHARACTERISTICS:
Population: Baseline population included all randomized participants who received study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sirukumab 50 Milligram (mg) | Sirukumab 100 mg | Total
Number analyzed (Participants) | 61 | 61 | 122
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (10.7) | 54.7 (12.16) | 55.1 (11.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 43 | 90
  Male | 14 | 18 | 32
Region of Enrollment [Number; unit: participants]
  JAPAN | 61 | 61 | 122

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAE)
Description: A TEAE was defined as an event that occurred in the treatment period during which it emerged (that is [i.e.] started or worsened in severity, relation, or other attribute), and even if the event continued to be present.
Time Frame: Baseline upto Week 68
Population: Safety analyses set included all participants who received at least 1 (partial or complete) dose of the study drug.
Measure: Number; unit: participants
Arm/Group | Sirukumab 50 Milligram (mg) | Sirukumab 100 mg
Number analyzed (Participants) | 61 | 61
participants | 56 | 58

2. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology (ACR) 20 Response
Description: The ACR 20 Response is defined as greater than or equal to (>=) 20 percent improvement in swollen joint count (66 joints) and tender joint count (68 joints) and >=20 percent improvement in 3 of following 5 assessments: patient's assessment of pain using Visual Analog Scale (VAS; 0-10 millimeter [mm], 0 mm=no pain and 10 mm=worst possible pain), patient's global assessment of disease activity by using VAS (the scale ranges from 0 mm to 100 mm, [0 mm=no pain to 100 mm=worst possible pain]), physician's global assessment of disease activity using VAS, participant's assessment of physical function measured by Health Assessment Questionnaire-Disability Index (HAQ-DI, defined as a 20-question instrument assessing 8 functional areas. The derived HAQ-DI ranges from 0, indicating no difficulty, to 3, indicating inability to perform a task in that area) and serum C-Reactive Protein (CRP).
Time Frame: At Weeks 16 and 24
Population: All participants randomly assigned to a treatment group were included in the efficacy analysis regardless of whether they received the assigned treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Sirukumab 50 Milligram (mg) | Sirukumab 100 mg
Number analyzed (Participants) | 61 | 61
percentage of participants
  Week 16 | 77.0 | 72.1
  Week 24 | 73.8 | 82.0

3. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology (ACR) 50 Response
Description: The ACR 50 Response is defined as >=50 percent improvement in swollen joint count (66 joints) and tender joint count (68 joints) and >=50 percent improvement in 3 of following 5 assessments: patient's assessment of pain using VAS (0-10 mm, 0 mm=no pain and 10 mm=worst possible pain), patient's global assessment of disease activity by using VAS (the scale ranges from 0 mm to 100 mm, [0 mm=no pain to 100 mm=worst possible pain]), physician's global assessment of disease activity using VAS, participant's assessment of physical function measured by HAQ-DI and serum CRP.
Time Frame: At Weeks 16 and 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Sirukumab 50 Milligram (mg) | Sirukumab 100 mg
Number analyzed (Participants) | 61 | 61
percentage of participants
  Week 16 | 47.5 | 57.4
  Week 24 | 49.2 | 63.9

4. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology (ACR) 70 Response
Description: The ACR 70 Response is defined as >=70 percent improvement in swollen joint count (66 joints) and tender joint count (68 joints) and >=70 percent improvement in 3 of following 5 assessments: patient's assessment of pain using VAS (0-10 mm, 0 mm=no pain and 10 mm=worst possible pain), patient's global assessment of disease activity by using VAS (the scale ranges from 0 mm to 100 mm, [0 mm=no pain to 100 mm=worst possible pain]), physician's global assessment of disease activity using VAS, participant's assessment of physical function measured by HAQ-DI and CRP.
Time Frame: At Weeks 16 and 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Sirukumab 50 Milligram (mg) | Sirukumab 100 mg
Number analyzed (Participants) | 61 | 61
percentage of participants
  Week 16 | 26.2 | 32.8
  Week 24 | 24.6 | 36.1

5. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology (ACR) 90 Response
Description: The ACR 90 Response is defined as >=90 percent improvement in swollen joint count (66 joints) and tender joint count (68 joints) and >=90 percent improvement in 3 of following 5 assessments: patient's assessment of pain using VAS (0-10 mm, 0 mm=no pain and 10 mm=worst possible pain), patient's global assessment of disease activity by using VAS (the scale ranges from 0 mm to 100 mm, [0 mm=no pain to 100 mm=worst possible pain]), physician's global assessment of disease activity using VAS, participant's assessment of physical function measured by HAQ-DI and CRP.
Time Frame: At Weeks 16 and 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Sirukumab 50 Milligram (mg) | Sirukumab 100 mg
Number analyzed (Participants) | 61 | 61
percentage of participants
  Week 16 | 8.2 | 11.5
  Week 24 | 6.6 | 14.8

6. Secondary Outcome: Percent Change From Baseline in Number of Swollen Joints at Weeks 16 and 24
Description: Sixty six (66) joints were assessed for swelling by investigator to determine the number of joints that were considered swollen. A negative change from baseline in swollen joint count indicates improvement.
Time Frame: Baseline, Weeks 16 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Sirukumab 50 Milligram (mg) | Sirukumab 100 mg
Number analyzed (Participants) | 61 | 61
percent change
  Change at Week 16 | -65.66 (40.201) | -73.84 (31.162)
  Change at Week 24 | -71.16 (38.343) | -75.82 (30.860)

7. Secondary Outcome: Percent Change From Baseline in Number of Tender Joints at Weeks 16 and 24
Description: Sixty eight (68) joints were assessed for tenderness to determine the number of joints that were considered tender. A negative change from baseline in the tender joint count indicates improvement.
Time Frame: Baseline, Weeks 16 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Sirukumab 50 Milligram (mg) | Sirukumab 100 mg
Number analyzed (Participants) | 61 | 61
percent change
  Change at Week 16 | -63.95 (41.738) | -65.58 (41.898)
  Change at Week 24 | -65.58 (41.933) | -67.34 (42.145)

8. Secondary Outcome: Percent Change From Baseline in Patient's Assessment of Pain at Weeks 16 and 24
Description: Participants assessed their average pain during the past week on a visual analogue scale (VAS). The scale ranged from 0 (no pain) to 10 (the worst possible pain).
Time Frame: Baseline, Weeks 16 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Sirukumab 50 Milligram (mg) | Sirukumab 100 mg
Number analyzed (Participants) | 61 | 61
percent change
  Change at Week 16 | -53.44 (39.043) | -52.94 (44.384)
  Change at Week 24 | -52.45 (38.266) | -57.56 (49.725)

9. Secondary Outcome: Percent Change From Baseline in Patient's Global Assessment of Disease Activity at Weeks 16 and 24
Description: Participants rated their disease activity using the Visual Analog Scale (VAS) on a scale of 0 (very well) to 10 (very poor).
Time Frame: Baseline, Weeks 16 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Sirukumab 50 Milligram (mg) | Sirukumab 100 mg
Number analyzed (Participants) | 61 | 61
percent change
  Change at Week 16 | -50.64 (48.679) | -53.15 (38.925)
  Change at Week 24 | -51.55 (50.569) | -56.94 (42.208)

10. Secondary Outcome: Percent Change From Baseline in Physician's Global Assessment of Disease Activity at Weeks 16 and 24
Description: Physician's Global Assessment of Disease Activity was assessed using the VAS on a scale of 0 (no arthritis activity) to 10 (extremely active arthritis).
Time Frame: Baseline, Weeks 16 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Sirukumab 50 Milligram (mg) | Sirukumab 100 mg
Number analyzed (Participants) | 61 | 61
percent change
  Change at Week 16 | -65.28 (27.268) | -66.17 (28.774)
  Change at Week 24 | -67.54 (25.521) | -68.44 (27.161)

11. Secondary Outcome: Percent Change From Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) at Weeks 16 and 24
Description: The HAQ-DI is a 20-question instrument that assesses the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping and activities of daily living). Responses in each functional area are scored from 0 to 3 (0=no difficulty and 3=inability to perform a task in that area). Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0 = least difficulty and 3 = extreme difficulty. Here, 'n' signifies those participants who were evaluable for the specific timepoint.
Time Frame: Baseline, Weeks 16 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Sirukumab 50 Milligram (mg) | Sirukumab 100 mg
Number analyzed (Participants) | 61 | 61
percent change
  Change at Week 16 (n= 59, 58) | -38.90 (53.204) | -46.18 (48.572)
  Change at Week 24 (n= 59, 58) | -42.25 (52.741) | -48.98 (44.917)

12. Secondary Outcome: Percent Change From Baseline in C-Reactive Protein (CRP) at Weeks 16 and 24
Description: Serum CRP is a marker of systemic inflammation. A negative percent change from baseline in CRP represents improvement.
Time Frame: Baseline, Weeks 16 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Sirukumab 50 Milligram (mg) | Sirukumab 100 mg
Number analyzed (Participants) | 61 | 61
percent change
  Change at Week 16 | -98.60 (2.026) | -98.97 (1.637)
  Change at Week 24 | -98.64 (2.148) | -98.99 (1.251)

13. Secondary Outcome: Percentage of Participants Who Achieved Major Clinical Response at Week 52
Description: Major clinical response is achieving ACR 70 for 6 continuous months. The ACR 70 Response is defined as >=70 percent improvement in swollen joint count (66 joints) and tender joint count (68 joints) and >=70 percent improvement in 3 of following 5 assessments: patient's assessment of pain using VAS (0-10 mm, 0 mm=no pain and 10 mm=worst possible pain), patient's global assessment of disease activity by using VAS, (The scale ranges from 0 mm to 100 mm, [0 mm=no pain to 100 mm=worst possible pain]), physician's global assessment of disease activity using VAS, participant's assessment of physical function measured by HAQ-DI and CRP. Achievement of major clinical response reflects an enhanced level of therapeutic efficacy and sustained reduction of signs and symptoms of rheumatoid arthritis (RA).
Time Frame: Week 52
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Sirukumab 50 Milligram (mg) | Sirukumab 100 mg
Number analyzed (Participants) | 61 | 61
percentage of participants | 13.1 | 24.6

14. Secondary Outcome: Percentage of Participants With Disease Activity Index Score 28 (CRP) Response at Weeks 16 and 24
Description: The DAS28 based on C-Reactive Protein (CRP) is a statistically derived index combining tender joints (28 joints), swollen joints (28 joints), CRP and patient's global assessment of disease activity. The set of 28 joint count is based on evaluation of the shoulder, elbow, wrist, metacarpophalangeal (MCP) MCP1 to MCP5, proximal interphalangeal (PIP) PIP1 to PIP5 joints of both the upper right extremity and the upper left extremity as well as the knee joints of lower right and lower left extremities. The values are 0=best to 10=worst. Good responders: improvement from baseline greater than (>) 1.2 with DAS28 less than or equal to (<=) 3.2; moderate responders: improvement from baseline >1.2 with DAS28 >3.2 to <=5.1 or improvement from baseline >0.6 to <=1.2 with DAS28 <=5.1; non-responders: improvement from baseline <=0.6 or improvement from baseline >0.6 and <=1.2 with DAS28 >5.1.
Time Frame: At Weeks 16 and 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Sirukumab 50 Milligram (mg) | Sirukumab 100 mg
Number analyzed (Participants) | 61 | 61
percentage of participants
  Week 16 | 90.2 | 96.7
  Week 24 | 88.5 | 96.7

15. Secondary Outcome: Percentage of Participants Achieving DAS28 (CRP) Remission at Week 24
Description: The DAS28 based on C-Reactive Protein (CRP) is a statistically derived index combining tender joints (28 joints), swollen joints (28 joints), CRP and patient's global assessment of disease activity. The set of 28 joint count is based on evaluation of the shoulder, elbow, wrist, metacarpophalangeal (MCP) MCP1 to MCP5, proximal interphalangeal (PIP) PIP1 to PIP5 joints of both the upper right extremity and the upper left extremity as well as the knee joints of lower right and lower left extremities. DAS28 (CRP) remission is defined as a DAS28 (CRP) value of less than (<) 2.6 at any study visit.
Time Frame: At Week 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Sirukumab 50 Milligram (mg) | Sirukumab 100 mg
Number analyzed (Participants) | 61 | 61
percentage of participants | 49.2 | 59.0

16. Secondary Outcome: Change From Baseline in DAS28 (CRP) Score at Weeks 16 and 24
Description: The DAS28 based on C-Reactive Protein (CRP) is a statistically derived index combining tender joints (28 joints), swollen joints (28 joints), CRP and patient's global assessment of disease activity. The set of 28 joint count is based on evaluation of the shoulder, elbow, wrist, metacarpophalangeal (MCP) MCP1 to MCP5, proximal interphalangeal (PIP) PIP1 to PIP5 joints of both the upper right extremity and the upper left extremity as well as the knee joints of lower right and lower left extremities. The values are 0=best to 10=worst.
Time Frame: Baseline, Weeks 16 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sirukumab 50 Milligram (mg) | Sirukumab 100 mg
Number analyzed (Participants) | 61 | 61
units on a scale
  Baseline | 5.566 (0.8088) | 5.805 (1.0553)
  Change at Week 16 | -2.858 (1.1867) | -3.069 (1.1483)
  Change at Week 24 | -2.949 (1.2445) | -3.185 (1.1552)

17. Secondary Outcome: Percentage of Participants With Simplified Disease Activity Index (SDAI) Based ACR/European League Against Rheumatism (EULAR) Remission at Weeks 16, 24 and 52
Description: The SDAI score is a derived score combining tender joints (28 joints), swollen joints (28 joints), patient's global assessment of disease activity on VAS, physician's global assessments of disease activity on VAS, and CRP. SDAI-based ACR/EULAR remission is defined as a SDAI value of <=3.3 at the visit.
Time Frame: At Weeks 16, 24 and 52
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Sirukumab 50 Milligram (mg) | Sirukumab 100 mg
Number analyzed (Participants) | 61 | 61
percentage of participants
  Week 16 | 14.8 | 19.7
  Week 24 | 16.4 | 18.0
  Week 52 | 18.0 | 26.2

18. Secondary Outcome: Percentage of Participants With Boolean Based ACR/EULAR Remission at Weeks 16, 24 and 52
Description: The Boolean based ACR/EULAR remission is achieved if all of the following 4 criteria at that visit are met: tender joint count (68 joints) <=1; swollen joint count (66 joints) <=1; CRP <=1 milligram per deciliter (mg/dL); and patient's global assessment of disease activity on visual analog scale (VAS) <=1 on a 0 to 10 scale.
Time Frame: At Weeks 16, 24 and 52
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Sirukumab 50 Milligram (mg) | Sirukumab 100 mg
Number analyzed (Participants) | 61 | 61
percentage of participants
  Week 16 | 4.9 | 14.8
  Week 24 | 9.8 | 8.2
  Week 52 | 8.2 | 13.1

19. Secondary Outcome: Change From Baseline in Clinical Disease Activity Index (CDAI) Score at Weeks 16 and 24
Description: The CDAI score is a derived score combining tender joints (28 joints), swollen joints (28 joints), patient's global assessment of disease activity, and physician's global assessments of disease activity. The total score range is 0-76. Score interpretation: Remission <=2.8; Low Disease Activity CDAI > 2.8 and <=10; Moderate Disease Activity CDAI >10 and <=22; High Disease Activity CDAI > 22.
Time Frame: Baseline, Weeks 16 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sirukumab 50 Milligram (mg) | Sirukumab 100 mg
Number analyzed (Participants) | 61 | 61
units on a scale
  Baseline | 31.36 (9.454) | 35.69 (13.923)
  Change at Week 16 | -19.43 (12.138) | -22.69 (13.231)
  Change at Week 24 | -20.27 (12.207) | -23.86 (13.487)

20. Secondary Outcome: Change From Baseline in Simplified Disease Activity Index (SDAI) Score at Weeks 16 and 24
Description: The SDAI score is a derived score combining tender joints (28 joints), swollen joints (28 joints), patient's global assessment of disease activity, physician's global assessments of disease activity, and CRP. The total score range is 0-86. Score interpretation: Remission SDAI <=3.3; Low Disease Activity SDAI >3.3 and <=11; Moderate Disease Activity SDAI >11 and <=26; High Disease Activity SDAI >26.
Time Frame: Baseline, Weeks 16 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sirukumab 50 Milligram (mg) | Sirukumab 100 mg
Number analyzed (Participants) | 61 | 61
units on a scale
  Baseline | 34.318 (9.6078) | 38.911 (14.7996)
  Change at Week 16 | -22.365 (12.4411) | -25.896 (13.9910)
  Change at Week 24 | -23.206 (12.6842) | -27.064 (14.2368)

21. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) Score at Week 16 and 24
Description: The HAQ-DI is a 20-question instrument that assesses the degree of difficulty a participant has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and activities of daily living), each scored from 0 (no difficulty) to 3 (inability to perform a task in that area). Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0 = least difficulty and 3 = extreme difficulty.
Time Frame: Baseline, at Week 16 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sirukumab 50 Milligram (mg) | Sirukumab 100 mg
Number analyzed (Participants) | 61 | 61
units on a scale
  Baseline | 1.3484 (0.65396) | 1.1721 (0.64111)
  Change at Week 16 | -0.5676 (0.53695) | -0.4980 (0.61343)
  Change at Week 24 | -0.5738 (0.54600) | -0.5697 (0.56758)

22. Secondary Outcome: Percentage of Participants Achieving HAQ-DI Response at Weeks 16 and 24
Description: The HAQ-DI is a 20-question instrument that assesses the degree of difficulty a participant has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and activities of daily living), each scored from 0 (no difficulty) to 3 (inability to perform a task in that area). HAQ-DI response was defined as change of > -0.22 from baseline in HAQ-DI score.
Time Frame: At Weeks 16 and 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Sirukumab 50 Milligram (mg) | Sirukumab 100 mg
Number analyzed (Participants) | 61 | 61
percentage of participants
  Week 16 | 75.4 | 67.2
  Week 24 | 73.8 | 70.5

23. Secondary Outcome: Percentage of Participants Maintaining HAQ-DI Response
Description: The HAQ-DI is a 20-question instrument that assesses the degree of difficulty a participant has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and activities of daily living), each scored from 0 (no difficulty) to 3 (inability to perform a task in that area). HAQ-DI responders who maintain a change from baseline of > -0.22 in HAQ-DI score.
Time Frame: Baseline upto Week 52
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Sirukumab 50 Milligram (mg) | Sirukumab 100 mg
Number analyzed (Participants) | 61 | 61
percentage of participants | 70.5 | 65.6

24. Secondary Outcome: Area Under Curve (AUC) of Change From Baseline in HAQ-DI Score From Week 0 Through Week 24 and From Week 0 Through Week 52
Description: HAQ-DI consisted of 20-question in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and activities of daily living), each scored from 0 (no difficulty) to 3 (inability to perform a task in that area). Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0 = least difficulty and 3 = extreme difficulty. AUC of change from baseline in HAQ-DI score is the AUC of change from baseline in HAQ-DI score versus the time. AUC was calculated based on the measurement (i.e., observed HAQ-DI score change from baseline) at scheduled visits using the trapezoidal rule. Functional status was determined as a cumulative measure of HAQ-DI over 1 year by using the AUC of the change from baseline in HAQ-DI score through week 52. Decreases in AUC of change from baseline in HAQ-DI indicate a greater average improvement in physical function over time.
Time Frame: Baseline, Weeks 24 and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale*week
Arm/Group | Sirukumab 50 Milligram (mg) | Sirukumab 100 mg
Number analyzed (Participants) | 61 | 61
units on a scale*week
  Week 0 Through Week 24 | -74.0645 (78.34712) | -69.2439 (75.85153)
  Week 0 Through Week 52 | -189.2531 (178.07291) | -187.4068 (191.77329)

25. Secondary Outcome: Change From Baseline in Duration of Morning Stiffness at Weeks 16 and 24
Description: Duration of morning stiffness was defined as the time elapsed when participant woke up in the morning and was able to resume normal activities without stiffness in minutes (If none was present = 0; If morning stiffness was continuing at the time of assessment or was unusual compared to the recent past, average of duration of stiffness over the past 3 days was reported; If stiffness persisted the entire day, 1440 minutes was recorded). Negative values for this outcome measure represent improvement, i.e. shortening of duration of morning stiffness.
Time Frame: Baseline, Weeks 16 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: minute
Arm/Group | Sirukumab 50 Milligram (mg) | Sirukumab 100 mg
Number analyzed (Participants) | 61 | 61
minute
  Change at Week 16 | -103.8 (268.32) | -160.4 (374.17)
  Change at Week 24 | -77.6 (334.00) | -169.4 (374.36)

26. Secondary Outcome: Change From Baseline in Mental Component Scores of 36-Item Short Form Health Survey (SF-36) at Weeks 16, 24 and 52
Description: The SF-36 is a survey of participant health. It consists of 8 individual domains, which are weighted sums of the questions in their section. The 8 domains are: vitality (VT), physical functioning (PF), bodily pain (BP), general health (GH), Role-Physical (RP), Role-Emotional (RE), social functioning (SF) and mental health (MH). Each of these 8 scales (domains) is scored from 0 to 100 with higher scores indicating better health. Based on the scale scores, the summary mental component score (MCS) is derived. Scales contributing most to the scoring of the SF-36 MCS include the VT, SF, RE and MH. Other domains not noted contribute to the scoring but to a lesser degree. The scoring is derived based on an algorithm that has been developed in a software provided by the developer. The summary MCS score is also scaled from 0 to 100 with higher scores indicating better health.
Time Frame: Baseline, Weeks 16, 24 and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sirukumab 50 Milligram (mg) | Sirukumab 100 mg
Number analyzed (Participants) | 61 | 61
units on a scale
  Baseline (Mental Component Score [MCS]) | 45.49 (9.577) | 46.55 (11.332)
  Change at Week 16 (MCS) | 5.38 (9.655) | 6.46 (9.183)
  Change at Week 24 (MCS) | 5.82 (10.376) | 6.81 (9.273)
  Change at Week 52 (MCS) | 6.74 (9.681) | 6.27 (9.915)

27. Secondary Outcome: Change From Baseline in Physical Component Scores of 36-Item Short Form Health Survey (SF-36) at Weeks 16, 24 and 52
Description: The SF-36 is a survey of participant health. It consists of 8 individual domains, which are weighted sums of the questions in their section. The 8 domains are: vitality (VT), physical functioning (PF), bodily pain (BP), general health (GH), Role-Physical (RP), Role-Emotional (RE), social functioning (SF) and mental health (MH). Each of these 8 scales (domains) is scored from 0 to 100 with higher scores indicating better health. Based on the scale scores, the summary physical component score (PCS) is derived. Scales contributing most to the scoring of the SF-36 PCS include the PF, RP, BP and GH. Other domains not noted contribute to the scoring but to a lesser degree. The scoring is derived based on an algorithm that has been developed in a software provided by the developer. The summary PCS score is also scaled from 0 to 100 with higher scores indicating better health.
Time Frame: Baseline, Weeks 16, 24 and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sirukumab 50 Milligram (mg) | Sirukumab 100 mg
Number analyzed (Participants) | 61 | 61
units on a scale
  Baseline (Physical Component Score [PCS]) | 22.12 (15.315) | 24.10 (15.642)
  Change at Week 16 (PCS) | 12.12 (14.349) | 12.48 (15.886)
  Change at Week 24 (PCS) | 12.45 (15.979) | 14.72 (15.290)
  Change at Week 52 (PCS) | 13.67 (15.754) | 14.30 (15.395)

28. Secondary Outcome: Change From Baseline in EuroQol 5-Dimensional Questionnaire (EQ-5D) Visual Analog Scale (VAS) Score at Weeks 16, 24 and 52
Description: The EQ-5D VAS records the participant's self-rated health on a vertical, VAS, with 0 representing the worst imaginable health state and 100 representing the best imaginable health state. The EQ VAS is used as a quantitative measure of health outcome as judged by the individual participant.
Time Frame: Baseline, Weeks 16, 24 and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sirukumab 50 Milligram (mg) | Sirukumab 100 mg
Number analyzed (Participants) | 61 | 61
units on a scale
  Change at Week 16 | 30.20 (26.145) | 25.93 (27.371)
  Change at Week 24 | 32.46 (26.562) | 28.85 (28.397)
  Change at Week 52 | 33.54 (26.972) | 31.50 (29.666)

29. Secondary Outcome: Change From Baseline in EuroQol 5-Dimensional Questionnaire (EQ-5D) Index Score at Weeks 16, 24 and 52
Description: Change from Baseline to end point in Euro Quality of life (Qol)-5 Dimension Questionnaire (EQ-5D). A higher score indicates an improvement in health in the Health Status Index. The EuroQol-5 is a five dimensional health state classification. Each dimension is assessed on a 3-point ordinal scale (1=no problems, 2=some problems, 3=extreme problems). The responses to the five EQ-5D dimensions were scored using a utility-weighted algorithm to derive an EQ-5D health status index score between 0 to 1, with 1.00 indicating "full health" and 0 representing dead.
Time Frame: Baseline, Weeks 16, 24 and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sirukumab 50 Milligram (mg) | Sirukumab 100 mg
Number analyzed (Participants) | 61 | 61
units on a scale
  Change at Week 16 | 0.16 (0.173) | 0.18 (0.177)
  Change at Week 24 | 0.17 (0.169) | 0.19 (0.172)
  Change at Week 52 | 0.16 (0.164) | 0.19 (0.166)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 68
Arm/Group | Sirukumab 50 Milligram (mg) | Sirukumab 100 mg
Serious Adverse Events (participants affected / at risk) | 4/61 | 5/61
Other Adverse Events (participants affected / at risk) | 48/61 | 51/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sirukumab 50 Milligram (mg) (N=61) | Sirukumab 100 mg (N=61)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 1
Large Intestine Polyp (Gastrointestinal disorders) | 1 | 0
Acute Sinusitis (Infections and infestations) | 0 | 1
Hepatitis E (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 1 | 0
Comminuted Fracture (Injury, poisoning and procedural complications) | 1 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Borderline Serous Tumour of Ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Schizophrenia (Psychiatric disorders) | 1 | 0
Endometriosis (Reproductive system and breast disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sirukumab 50 Milligram (mg) (N=61) | Sirukumab 100 mg (N=61)
Diarrhoea (Gastrointestinal disorders) | 5 | 3
Injection Site Erythema (General disorders) | 19 | 20
Injection Site Pruritus (General disorders) | 7 | 13
Injection Site Swelling (General disorders) | 10 | 12
Bronchitis (Infections and infestations) | 5 | 0
Gastroenteritis (Infections and infestations) | 4 | 1
Nasopharyngitis (Infections and infestations) | 27 | 27
Paronychia (Infections and infestations) | 6 | 2
Pharyngitis (Infections and infestations) | 6 | 7
Tinea Pedis (Infections and infestations) | 4 | 1
Skin Abrasion (Injury, poisoning and procedural complications) | 4 | 1
Alanine Aminotransferase Increased (Investigations) | 10 | 10
Aspartate Aminotransferase Increased (Investigations) | 9 | 11
Neutrophil Count Decreased (Investigations) | 7 | 4
Platelet Count Decreased (Investigations) | 9 | 3
White Blood Cell Count Decreased (Investigations) | 7 | 7
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 0 | 4
Eczema (Skin and subcutaneous tissue disorders) | 7 | 7
Rash (Skin and subcutaneous tissue disorders) | 1 | 4
Urticaria (Skin and subcutaneous tissue disorders) | 4 | 3
Hypertension (Vascular disorders) | 5 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.